CLINICAL TRIAL: NCT02664181
Title: Phase II Evaluation of Nivolumab, an Immune Checkpoint Inhibitor Alone or in Combination With Oral Decitabine/Tetrahydrouridine as Second Line Therapy for Non-small Cell Lung Cancer
Brief Title: Rational EpigenetiC Immunotherapy for SEcond Line Therapy in Patients With NSCLC: PRECISE Trial
Acronym: PRECISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yogen Saunthararajah, Professor of Medicine, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3516; NCT02795923 (obsolete NCT alias)
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: Cancer; Nivolumab; Decitabine; Tetrahydrouridine
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Nivolumab; Decitabine; Tetrahydrouridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral THU/decitabine + Nivolumab (Experimental): Oral THU ~10 mg/kg, followed by oral decitabine ~0.2 mg/kg 60 minutes after the THU, twice weekly on consecutive days. This drug combination is administered with Nivolumab 3mg/kg IV Q2 weeks until progression
  Interventions: Drug: Nivolumab; Drug: oral decitabine; Drug: Tetrahydrouridine
- Nivolumab (Active Comparator): Nivolumab 3mg/kg IV Q2 weeks until progression; This is the standard of care for patients with NSCLC who have progressed on prior chemotherapy.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given at 3mg/kg by IV every two weeks until progression
  Other Names: Opdivo
Drug: oral decitabine — oral decitabine ~0.2 mg/kg 60 minutes after the THU, twice weekly on consecutive days.
  Other Names: decitabine; DEC; Dacogen
  Arms: Oral THU/decitabine + Nivolumab
Drug: Tetrahydrouridine — Oral THU ~10 mg/kg twice weekly on consecutive days
  Other Names: THU
  Arms: Oral THU/decitabine + Nivolumab

SUMMARY:
The purpose of this study is to assess whether treatment with the study drug tetrahydrouridine-decitabine (THU-Dec) in combination with nivolumab is more effective than treatment with nivolumab alone in patients with NSCLC.

Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1 (DNMT1). DNMT1 is an enzyme, or protein that causes chemical changes, often increased in cancer. Blocking DNMT1 has been shown to reduce tumor formation. Decitabine is experimental in this study because it is not approved by the Food and Drug Administration (FDA) for patients with lung cancer. Decitabine is approved by the FDA for treating patients with a blood disease called myelodysplastic syndrome (MDS, a condition where the bone marrow does not make blood cells normally).

THU is an investigational (experimental) drug that works by blocking an enzyme that breaks down decitabine. This enzyme is highly expressed in solid tissues of the body, limiting the distribution of decitabine into these tissues, including solid cancer tissues. So, THU will increase the time cells are exposed to decitabine. The idea is that THU will also increase the time that the lung cancer cells are exposed to decitabine. THU is experimental because it is also not approved by the FDA, although it has been extensively used in clinical trials, including several cancer trials.

DETAILED DESCRIPTION:
Primary objective: To determine if non-cytotoxic oral THU-Dec when combined with nivolumab can improve objective response rates of nivolumab

Secondary objectives:

i) To evaluate clinical efficacy end points and toxicity of oral THU-Dec when combined with nivolumab ii) evaluate the induction of a T-cell response in patients with metastatic NSCLC iii) To evaluate hypotheses regarding mechanisms of resistance and predictive biomarkers for response to nivolumab

Study design: This is a Phase 2 randomized two arm trial of nivolumab alone or in combination with THU-Dec, in previously treated patients with stage IV Non-Small Cell Lung Cancer (NSCLC). The primary goal of this trial is to compare the efficacy of oral THU-Dec as a way of enhancing the anti-tumor immune response to nivolumab to that of nivolumab alone. The primary efficacy endpoint is overall RECIST-defined response. To accomplish this goal 60 patients will be randomized 2:1 to THU-Dec plus nivolumab or nivolumab only respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven NSCLC
* Subjects must have received 1 or more prior systemic therapies for this disease, should not have had prior treatment with immunotherapy; (including immune checkpoint inhibitor drugs, or immunotherapy vaccines); Patients with epidermal growth factor receptor (EGFR) or ALK alterations will need to have progressed on a TKI treatment
* Measurable disease per RECIST1.1
* Disease that can be accessed by a bronchoscopic, surgical or percutaneous biopsy

  * Eligible for biopsy from safety perspective
  * Agrees to percutaneous biopsy prior to study, may be eligible if archival tissue from a biopsy is after most recent therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Adequate organ function as defined by the following criteria:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥8.5g/dL or ≥5.6mmol/L
  * Serum creatinine ≤1.5 times upper limit of normal
  * Measured or calculated creatinine clearance ≥ 30mL/min for subject with creatinine levels > 1.5 times institutional upper level of normal (ULN)
  * Serum total bilirubin ≤1.5 times upper limit of normal
  * Direct bilirubin ≤ upper limit of normal for subjects with total bilirubin levels > 1.5 upper limit of normal
  * AST (SGOT) ≤2.5 times upper limit of normal or ≤5 times upper limit of normal for subjects with liver metastases
  * ALT (SGPT) ≤2.5 times upper limit of normal or ≤5 times upper limit of normal for subjects with liver metastases
  * Albumin ≥ 2 mg/dL
* Patients with history of brain metastases can be eligible for study treatment at a minimum of 1 weeks following the completion of gamma knife or whole brain radiotherapy. (if patient underwent surgical resection of brain metastasis need to wait for 4 weeks before study treatment) Patients should ideally be off steroids at the start of study treatment, however patients on steroid taper and dose of no more than 2mg/day of Decadron at the time of study treatment are allowed; and steroids should be tapered off as quickly as clinically feasible.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass graft, New York Heart Association grade II or greater congestive heart failure, cerebrovascular accident or transient ischemic attack, clinically unstable bleeding or pulmonary embolism leading to hemodynamic compromise are not allowed
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with oral THU-Dec. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Pregnancy or breastfeeding (pregnant or breastfeeding women are excluded from this study because oral THU-Dec has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with oral THU-Dec, breastfeeding should be discontinued if the mother is treated with oral THU-Dec.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent; Patients who receive palliative radiation therapy within 1 week prior to day 1 are allowed. Patients on treatment with targeted therapy (like EGFR or ALK TKIs) may start study treatment 5 days from last treatment.
* Receiving other investigational agent
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin,in situ cervical cancer, superficial bladder cancer or localized low grade prostate cancer not requiring active treatment
* Has active and documented history of autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).Patients with psoriasis and rheumatoid arthritis with no evidence of disease flare off immunosuppression for >1year may be allowed after discussion with the study PI. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 217 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2024-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD,PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Center for Cancer Research, Bethesda, Maryland
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral THU/Decitabine + Nivolumab | Nivolumab
Started | 8 | 5
Completed | 8 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral THU/Decitabine + Nivolumab | Nivolumab | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Customized [Count of Participants; unit: Participants]
  years: 40-49 | 2 | 0 | 2
  years: 50-59 | 1 | 2 | 3
  years: 60-69 | 3 | 2 | 5
  years: 70-79 | 2 | 0 | 2
  years: 80-89 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response by Response Evaluation Criteria in Solid Tumors (RECIST1.1)
Description: Overall response rate (ORR) is defined as the proportion of all randomized subjects whose best overall response (BOR) from baseline is either a complete response (CR) or partial response (PR) per RECIST 1.1 criteria. BOR is determined by the best response designation recorded between the date of randomization and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. For subjects without documented progression or subsequent anticancer therapy, all available response designations will contribute to the BOR determination. For subjects who continue treatment beyond progression, the BOR should be determined based on response designations recorded at the time of the initial RECIST 1.1 defined progression.
Time Frame: Up to 52 weeks after beginning therapy
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Oral THU/Decitabine + Nivolumab
Number analyzed (Participants) | 5 | 8
Participants
  Progressive disease | 1 | 4
  Stable Disease | 3 | 2
  Partial Remission | 1 | 2
Statistical Analysis 1: Comparison: Nivolumab vs Oral THU/Decitabine + Nivolumab; Partial remission rate was compared between both arms. The null hypothesis is that there is no difference in partial remission rate between the two arms, with a p-value of < 0.05 indicating significance; Test type: Superiority; p = 0.05, Fisher Exact

2. Secondary Outcome: Time-to-Progression
Description: Time-to-Progression defined as the time from randomization to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause. Subjects who die without a reported prior progression will be considered to have progressed on the date of their death. Subjects who did not progress or die will be censored on the date of their last evaluable tumor assessment. Subjects who did not have any on study tumor assessments and did not die will be censored on the date they were randomized. Subjects who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last evaluable tumor assessment prior to initiation of the subsequent anti-cancer therapy. Progression will be assessed every 6 weeks (from the first on-study radiographic assessment) until disease progression is noted.
Time Frame: Up to 77 weeks after beginning treatment
Population: Participants enrolled in study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nivolumab | Oral THU/Decitabine + Nivolumab
Number analyzed (Participants) | 5 | 8
days | 227 [45 to 754] | 69 [19 to 399]
Statistical Analysis 1: Comparison: Nivolumab vs Oral THU/Decitabine + Nivolumab; Test type: Superiority; p = 0.06, Log Rank; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.13 to 1.21]

3. Secondary Outcome: Overall Survival
Description: Overall survival: It is defined as the time from randomization to the date of death. A subject who has not died will be censored at last known date alive. Overall survival (OS) will be followed continuously while subjects are on the study drug.
Time Frame: Up to 171 weeks after beginning treatment
Population: Participants enrolled in study
Measure: Median (Full Range); unit: Days
Arm/Group | Nivolumab | Oral THU/Decitabine + Nivolumab
Number analyzed (Participants) | 5 | 8
Days | 844 [127 to 1183] | 389.5 [36 to 1147]
Statistical Analysis 1: Comparison: Nivolumab vs Oral THU/Decitabine + Nivolumab; Test type: Superiority; p = 0.19, Log Rank; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.11 to 1.62] — Data from Kaplan-Meier analyses

4. Secondary Outcome: Overall Survival - Long Term Follow-up (LTFU)
Description: Survival LTFU is planned to be done until death or withdrawal of consent, or until the final clinical trial report is published
Time Frame: Up to 5 years from end of treatment
Population: In the Nivolumab arm, 3 subjects did not meet the criteria for this outcome measure per protocol (received less than 12 doses). In the Oral THU/Decitabine + Nivolumab arm, 2 subjects id not meet the criteria for this outcome measure per protocol (received less than 12 doses).
Measure: Mean (Full Range); unit: months
Arm/Group | Nivolumab | Oral THU/Decitabine + Nivolumab
Number analyzed (Participants) | 2 | 6
months | 5 [3 to 7] | 6.8 [1 to 17]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while the participants were on treatment for up to 20 months
Arm/Group | Oral THU/Decitabine + Nivolumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 6/8 | 3/5
Serious Adverse Events (participants affected / at risk) | 4/8 | 1/5
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral THU/Decitabine + Nivolumab (N=8) | Nivolumab (N=5)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral THU/Decitabine + Nivolumab (N=8) | Nivolumab (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (14) | 1 (8)
Absolute lymphocyte decrease (Investigations) | 1 (5) | 0 (0)
Absolute neutrophil decrease (Investigations) | 1 (3) | 0 (0)
akathisa (Investigations) | 1 (2) | 0 (0)
Alanine aminotransferase elevated (Investigations) | 1 (2) | 0 (0)
alanine aminotransferase increased (Investigations) | 1 (1) | 1 (6)
Alkaline phosphatase increased (Investigations) | 3 (9) | 0 (0)
ALT increased- due to prednisone (Investigations) | 1 (4) | 0 (0)
anemia (Blood and lymphatic system disorders) | 6 (63) | 2 (194)
anorexia (Metabolism and nutrition disorders) | 3 (5) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (17) | 1 (6)
Aspartate aminotransferase elevated (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (14)
Aspartate phosphate increased (Investigations) | 0 (0) | 1 (4)
AST increased- due to prednisone (Investigations) | 1 (4) | 0 (0)
Back & Joint Cramp (General disorders) | 0 (0) | 1 (1)
Back/Shoulder pain (General disorders) | 0 (0) | 1 (1)
Bilateral hip pain (General disorders) | 0 (0) | 1 (1)
Body ache (General disorders) | 0 (0) | 1 (2)
BONE PAIN (left lateral rib) (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (7)
Chronic Back Pain (General disorders) | 0 (0) | 1 (1)
Cold (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (14) | 1 (4)
Cough/ drainage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (8)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (16) | 1 (6)
Dizziness (Nervous system disorders) | 2 (5) | 1 (149)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (7) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (8)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Edema limbs (General disorders) | 1 (1) | 2 (24)
Fatigue (General disorders) | 5 (29) | 1 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Hot & Cold sweats at night (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 2 (25) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (7) | 2 (19)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (13) | 2 (18)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (100)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Knee & Ankle Pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
lymphocyte count decreased (Investigations) | 3 (13) | 1 (1)
mucosal infection (Infections and infestations) | 1 (2) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (14) | 0 (0)
Nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (3)
Neck Pain (General disorders) | 0 (0) | 1 (1)
neutrophil count decreased (Investigations) | 3 (5) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
pain (left rib) (General disorders) | 1 (1) | 0 (0)
pain in extremity (left arm) (General disorders) | 0 (0) | 1 (18)
Pain, musculoskeletal, Left flank (General disorders) | 0 (0) | 1 (6)
papulopustular rash (Infections and infestations) | 1 (15) | 0 (0)
periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (100)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (15) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0)
Side Pain (General disorders) | 0 (0) | 1 (1)
skin infection - fungal rash around urostomy (Infections and infestations) | 1 (4) | 0 (0)
spasticity - left elbow (Nervous system disorders) | 1 (4) | 0 (0)
supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (156)
Upper respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0)
White blood cell decreased (Investigations) | 4 (18) | 0 (0)
worsening paraesthesia (Nervous system disorders) | 1 (4) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02664181/Prot_SAP_002.pdf
  • Informed Consent Form (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT02664181/ICF_001.pdf